CLINICAL TRIAL: NCT03559062
Title: A Phase 3, Double-blind, Parallel-group Study to Evaluate the Efficacy and Safety of Tezacaftor in Combination With Ivacaftor in Subjects Aged 6 Through 11 Years With Cystic Fibrosis, Homozygous or Heterozygous for the F508del-CFTR Mutation
Brief Title: A Study to Evaluate Efficacy and Safety of TEZ/IVA in Subjects Aged 6 Through 11 Years With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX16-661-115; 2016-004479-35 (EudraCT Number)
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Other): Participants with genotype F/F received placebo matched to TEZ/IVA fixed dose combination (FDC) in the morning and placebo matched to IVA in the evening for 8 weeks.
  Interventions: Drug: Placebo
- TEZ/IVA (Experimental): Participants with genotype F/F received TEZ/IVA FDC in the morning and IVA in the evening for 8 weeks. Participants with genotype F/RF received TEZ/IVA FDC and placebo matched to IVA in the morning and IVA in the evening for 8 weeks.
  Interventions: Drug: TEZ/IVA; Drug: IVA; Drug: Placebo
- Ivacaftor (Experimental): Participants with genotype F/RF received placebo matched to TEZ/IVA FDC in the morning and IVA in morning and evening for 8 weeks.
  Interventions: Drug: IVA; Drug: Placebo

INTERVENTIONS:
Drug: TEZ/IVA — Participants weighing <40 kg received TEZ 50 mg/IVA 75 mg FDC tablet and those weighing ≥40 kg received TEZ 100 mg/IVA 150 mg FDC tablet.
  Other Names: VX-661/VX-770; tezacaftor/ivacaftor fixed dose combination
  Arms: TEZ/IVA
Drug: IVA — Participants weighing <40 kg IVA 75 mg tablet and those weighing ≥40 kg received IVA 150 mg tablet.
  Other Names: VX-770; ivacaftor
  Arms: Ivacaftor; TEZ/IVA
Drug: Placebo — Placebo matched to TEZ/IVA FDC
  Arms: Ivacaftor; Placebo
Drug: Placebo — Placebo matched to IVA
  Arms: Placebo; TEZ/IVA

SUMMARY:
This study will evaluate the efficacy of tezacaftor in combination with ivacaftor (TEZ/IVA) in participants with cystic fibrosis (CF) aged 6 through 11 years, who are homozygous for the F508del mutation (F/F) or heterozygous for F508del with an eligible residual function mutation (F/RF).

ELIGIBILITY:
Key Inclusion Criteria:

* Homozygous for F508del or heterozygous for F508del and an RF mutation (as defined in the protocol).
* Participants with ppFEV1 of ≥70 percentage points adjusted for age, sex, height.
* Participants with a screening LCI2.5 result ≥7.5.
* Participants who are able to swallow tablets.

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension.
* Colonization with organisms associated with a more rapid decline in pulmonary status.
* Solid organ or hematological transplantation.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- Australia (4):
  - Hunter Medical Research Institute (HMRI), New Lambton Heights
  - Princess Margaret Hospital for Children, Perth
  - Lady Cilento Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- Belgium (2):
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- University of Copenhagen Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Groupe Hospitalier Pellegrin - Hôpital des Enfants, Bordeaux
  - Hôpital Necker - Enfants Malades, Paris
- Germany (8):
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Giessen, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Tuebingen, Tübingen
- Ireland (2):
  - Our Lady's Children's Hospital, Dublin
  - University Hospital Limerick, Limerick
- Klinika Mukowiscydozy, Oddział Chorób Płuc SZP ZOZ, Dziekanów Leśny, Poland
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Kinderspital Zuerich, Zurich
- United Kingdom (5):
  - Royal Hospital for Sick Children, Edinburgh
  - Leeds General Infirmary, Leeds
  - Royal Brompton Hospital, London
  - Nottingham University Hospital City Campus, Nottingham
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 69 participants were randomized, out of which 67 participants received study drug and were included in participant flow and baseline characteristics section.
Period: Overall Study
Arm/Group | Placebo | TEZ/IVA | Ivacaftor
Started | 10 | 54 | 3
Completed | 10 | 53 | 3
Not Completed | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TEZ/IVA | Ivacaftor | Total
Number analyzed (Participants) | 10 | 54 | 3 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.7) | 8.5 (1.7) | 9.0 (1.7) | 8.6 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 29 | 2 | 37
  Male | 4 | 25 | 1 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 46 | 3 | 59
  Unknown or Not Reported | 0 | 7 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 10 | 51 | 3 | 64
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Lung Clearance Index 2.5 (LCI2.5) [Mean (Standard Deviation); unit: lung clearance index] — LCI2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
  lung clearance index | 9.67 (1.65) | 9.56 (2.06) | 8.60 (1.40) | 9.54 (1.97)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Lung Clearance Index 2.5 (LCI2.5) Through Week 8
Description: LCI2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
Time Frame: From baseline through Week 8
Population: Full Analysis Set: all participants who were randomized, received at least 1 dose of study drug and had an eligible genotype. As per the pre-specified analysis, efficacy was only planned to be assessed for TEZ/IVA group. Placebo or IVA groups were used for blinding purposes only and were not applicable for the purpose of primary efficacy analysis.
Measure: Least Squares Mean (Standard Error); unit: lung clearance index
Arm/Group | TEZ/IVA
Number analyzed (Participants) | 54
lung clearance index | -0.51 (0.11)
Statistical Analysis 1: Comparison: TEZ/IVA; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure

2. Secondary Outcome: Absolute Change in Sweat Chloride At Week 8
Description: Sweat samples were collected using an approved collection device.
Time Frame: From baseline at Week 8
Population: FAS. As per the pre-specified analysis, efficacy was only planned to be assessed for TEZ/IVA group. Placebo or IVA groups were used for blinding purposes only and were not applicable for the purpose of secondary efficacy analysis.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | TEZ/IVA
Number analyzed (Participants) | 54
millimole per liter (mmol/L) | -12.3 (1.5)
Statistical Analysis 1: Comparison: TEZ/IVA; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure

3. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through Week 8
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From baseline through Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEZ/IVA
Number analyzed (Participants) | 54
units on a scale | 2.3 (1.2)
Statistical Analysis 1: Comparison: TEZ/IVA; Test type: Other; p = 0.0546, Mixed-effects model for repeated measure

4. Secondary Outcome: Safety and Tolerability as Assessed Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) up to Safety Follow-up Visit
Time Frame: From first dose of study drug up to safety follow-up visit (up to Week 12)
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEZ/IVA | Ivacaftor
Number analyzed (Participants) | 10 | 54 | 3
Participants
  Participants with AEs | 8 | 41 | 2
  Participants with SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to safety follow-up visit (up to Week 12)
Arm/Group | Placebo | TEZ/IVA | Ivacaftor
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/54 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/54 | 0/3
Other Adverse Events (participants affected / at risk) | 8/10 | 31/54 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | TEZ/IVA (N=54) | Ivacaftor (N=3)
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 8 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 3 | 0
Gastroenteritis (Infections and infestations) | 0 | 4 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 5 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT03559062/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT03559062/SAP_001.pdf